CLINICAL TRIAL: NCT00139646
Title: A Multicenter Single-Blind, Single Dose Efficacy and Safety Pilot Study Comparing Intramuscular Parecoxib and Diclofenac in Renal Colic
Brief Title: Parecoxib in Renal Colic
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 124-IFL-0505-005; A3481007
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Colic
MeSH Terms: conditions — Colic | interventions — parecoxib; Diclofenac

INTERVENTIONS:
Drug: Parecoxib
Drug: Diclofenac

SUMMARY:
This is a phase III, multicenter, randomized, single blind study designed to evaluate the efficacy and tolerability of a single dose of parecoxib compared with diclofenac in the treatment of acute pain due to renal colic.

DETAILED DESCRIPTION:
This study was prematurely discontinued May 3, 2004 due to slow recruitment. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of renal colic;
* baseline pain > 50 mm on VAS;

Exclusion Criteria:

* evidence of neoplasm or any other severe disease of any organ, including any psychiatric illness;
* active GI disease (e.g. Crohn's disease or ulcerative colitis) or any evidence of concomitant disease which may lead to early termination of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-04; Study Completion 2004-04

PRIMARY OUTCOMES:
Evaluation of efficacy through: time to onset of pain relief and time to remedication.

SECONDARY OUTCOMES:
Evaluation of efficacy through: Pain Intensity (VAS), Pain Relief (PR) and several measurements of analgesia that will be derived from VAS and PR Physician's Global Evaluation at 12 hours Patient's Global Evaluation at 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Italy (5):
  - Pfizer Investigational Site, Alessandria
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Siena

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=124-IFL-0505-005&StudyName=Parecoxib+in+renal+colic